CLINICAL TRIAL: NCT04820816
Title: Effect of Posterior Pelvic Tilt on Balance, Sensory Integration and Risk of Fall in Patients With Non-specific Low Back Pain
Brief Title: Effect of Posterior Pelvic Tilt on Balance and Sensory Integration in Patients With Non-specific Low Back Pain
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: MTI University (Other)
Responsible Party: Principal Investigator, Noha Abbas Abdelaziz Ali, Principle Investigator, MTI University
Other Study IDs: 012-003133
Record Dates: First submitted 2021-03-20; First posted 2021-03-29 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Biochemical Lesions Lumbar Region; Orthopedic Disorder of Spine; Back Disorder
Keywords: pelvic tilt; sensory integration; balance; back pain; biodex
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Posterior pelvic tilt group: 1. patients with chronic low back pain or repeated non-specific back pain for more than three months.
  2. Both sex with posterior pelvic tilt (-0.7 ± 6.5°) and decreased lumbar lordosis
  3. Their ages were ranged from 20-35 years
  4. Body Mass Index from 18-25 Kg/m²
  Interventions: Other: pelvic tilt effect on balance, sensory integration and risk of fall
- Normal anterior pelvic tilt group: 1. patients with chronic low back pain or repeated non-specific back pain for more than three months.
  2. Both sex with anterior pelvic tilt (5° and 13°) and normal lumbar lordosis
  3. Their ages were ranged from 20-35 years
  4. Body Mass Index from 18-25 Kg/m²
  Interventions: Other: pelvic tilt effect on balance, sensory integration and risk of fall

INTERVENTIONS:
Other: pelvic tilt effect on balance, sensory integration and risk of fall — BIODEX balance system, Limits of stability test, Risk of Fall test, m-CTSIB test

SUMMARY:
There is a debate in the literature about the effect of NSLBP on pelvic tilt and its effect on balance, sensory integration and functional disability so we need this study to fill the aforementioned gap in literature in this field. So the purpose of the study is to evaluate posterior pelvic tilt effect on overall dynamic balance, sensory integration and functional disability in patients with non-specific low back pain.

DETAILED DESCRIPTION:
The LBP became one of the biggest problems for public health systems in the world during the second half of the 20th century. The lifetime prevalence of LBP is reported to be as high as 84%, and the prevalence of chronic LBP is about 23%, with 11-12% of the population being disabled by LBP. Prevalence of LBP was 53.2%. It was more among female patients (62.8%) than among male patients (38.3%) among attendants to a Family Health Center in Egypt.

Additionally, studies have observed relationships between chronic non-specific LBP and a posteriorly shifted center of gravity, impaired proprioception, and decreased muscular strength, activation and endurance of the trunk and hips. Balance is impaired in individuals with chronic low back pain when compared to healthy individuals.

Most of these studies supposed that postural mal-alignment involves deviations in only one direction which is toward lordosis and anterior pelvic tilt. However, clinical experience suggests that some patients with back pain have the opposite problem which is a much reduced lordotic curve and a posterior pelvic tilt. If the true relationship between posture and low back pain disability is curvilinear instead, this could explain why the studies so far have shown weak or no relationships.

ELIGIBILITY:
Inclusion Criteria:

1. Fifty patients with chronic low back pain or repeated non-specific back pain for more than three months.
2. Both sex with posterior pelvic tilt (-0.7 ± 6.5°)and decreased lumbar lordosis, for (Group A) and normal anterior pelvic tilt angle between 5° and 13° for (Group B)
3. Their ages were ranged from 20-35 years.
4. Body Mass Index from 18-25 Kg/m² .

Exclusion Criteria:

1. Previous back surgery.
2. Signs and symptoms of gross spinal instability.
3. Radiological diagnosis of spondylolysis or spondylolisthesis.
4. Acute low back pain.
5. Disc prolapse or herniation.
6. Any neurological, orthopedic, and vestibular disorders affecting the balance system.
7. Flexion and extension restriction of the lumbar region.
8. Other conditions that affected the normal functioning of the central and peripheral nervous system such as alcohol abuse, addiction, dementia, and cognitive disorders.

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Fifty patients with chronic low back pain or repeated non-specific back pain for more than three months and referred from a physician with anterior or posterior pelvic tilt angles according to the groups.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-04-01 (Estimated); Study Completion 2021-04-15 (Estimated)

PRIMARY OUTCOMES:
Biodex balance system Limits of stability test | 10 minuets
  A test measures dynamic postural stability in percentage
Biodex balance system m-CTSIB test | 10 minuets
  A test measures postural sway control to assess sensory integration.
Biodex balance system Fall risk test (FR) | 10 minuets
  A test to assess risk of fall according to mean age
Oswestry Disability Index (ODI) | 10 minuets
  An index to assess physical functioning in percentage.

SECONDARY OUTCOMES:
The Global Posture System (GPS) 600 | 10 minuets
  A device to assess degree of pelvic tilt angle in degrees.
Body Mass Index (weight in kilograms, height in meters) | 10 minuets
  kg/m^2

CONTACTS AND LOCATIONS:
Overall Officials: Noha Abbas, MSc, Study Chair — MTI University
Locations (1):
- Noha Abbas Abdelaziz Ali, Cairo, Egypt